CLINICAL TRIAL: NCT01174043
Title: Pilot Study of Erlotinib for the Treatment of Patients With de Novo Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1006-12; IUCRO-0300
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Leukemia, Myelomonocytic, Acute
Keywords: Leukemia, Myelomonocytic, Acute; Erlotinib
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib will be administered orally at 150 mg once a day, continuously. Each cycle will be 28 days and there will be no break between the cycles.

SUMMARY:
This research study is looking for patients with newly diagnosed acute myeloid leukemia (AML), AML that has returned (relapsed), or it has not responded adequately to previous treatments. Treating certain patients with chemotherapy may not be to their benefit or may cause more harm than benefit. The purpose of this study is to find out what effects (good and bad) erlotinib has on patients and their AML.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML with no history of previous clonal/malignant hematologic disorders such as myelodysplastic syndromes or myeloproliferative disorders.
* Newly diagnosed patients will be age 70 or older
* Relapses patients will be age 60 or older any time following first relapse, if patient is not considered candidate/not interested in salvage chemotherapy.
* Refractory disease patients will be age 18-59 who have failed at least 2 lines of conventional chemotherapy (1 induction and 1 salvage)
* Patient must have discontinued all previous therapies for AML at least 14 days and recovered from the non-hematologic side effects of the therapy.
* Laboratory tests must be within protocol-specified ranges
* Patient must be able to swallow and tolerate oral medication.

Exclusion Criteria:

* Patients with known central nervous system (CNS) leukemia by spinal fluid cytology, flow cytometry or imaging.
* History of antecedent pre-leukemic hematologic disorders such as myelodysplastic syndromes or myeloproliferative disorders.
* Diagnosis of acute promyelocytic leukemia (APL)
* Patients who require chronic anticoagulation, are current smokers or who are taking rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital and St. John's Wort are not eligible.
* Patients with active corneal erosions or history of abnormal corneal sensitivity test.
* Patients with serious illness such as: significant ongoing or active infection, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable angina (anginal symptoms at rest), new onset angina (began within the last 3 months), myocardial infarction within the past 6 months, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy, cerebrovascular accident within past 3 months, or psychiatric illness that would limit compliance with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Hamid Sayar, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on getting 14 patients. Due to the lack of response, the study was stopped at 11 patients for this pilot study.
Period: Overall Study
Arm/Group | Erlotinib
Started | 11
Completed | 0
Not Completed | 11
Not completed — Disease progression | 5
Not completed — Adverse Event | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.8 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Defined as Partial Remission or Better) to 3 Months of Treatment With Erlotinib
Description: The percent of patients were shown as having a partial remission or better based on definitions of response in AML. Partial remission includes a decrease of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate. Complete remission includes presence of less than 5% blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. The percent and 95% exact confidence intervals will be calculated.
Time Frame: 3 months of treatment with erlotinib
Population: All patients enrolled and received treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
percentage of participants | 0 [0 to 0]

2. Secondary Outcome: Duration of Response (up to One Year Follow up) in Patients Who Achieve a Complete Remission
Description: The duration of response is from the time of response until failure or until the end of follow-up for the patients who received complete remission. Complete remission includes presence of less than 5% blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells.
Time Frame: 1 year after treatment discontinuation
Population: All patients enrolled and received treatment
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
months | 0 (0)

3. Secondary Outcome: Treatment Related Adverse Events Grade 3 or Higher
Description: Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Grading scale will be from 1 (mild) to 5 (causing death). This will determine the number of unique patients who had a treatment related (possible, probable or definite) adverse event that was graded 3 or greater.
Time Frame: up to 15 months
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
participants | 0

4. Other Pre Specified Outcome: Mechanistic Attributes of Erlotinib Hydrochloride in AML, Including Intracellular Quantitative Protein and Gene Expression Modifications and the in Vivo Effect of This Agent on the Differentiation of AML Blasts
Time Frame: Baseline; days 3, 4, 8, and 29 of course 1; and day 29 of courses 3, 6, 9, and 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=11)
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (Blood and lymphatic system disorders) | 2
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - ATRIAL FIBRILLATION (Cardiac disorders) | 1
DIARRHEA (Gastrointestinal disorders) | 2
HEPATOBILIARY/PANCREAS - OTHER (Hepatobiliary disorders) | 1
CREATININE (Investigations) | 1
SODIUM, SERUM-LOW (HYPONATREMIA) (Metabolism and nutrition disorders) | 1
URIC ACID, SERUM-HIGH (HYPERURICEMIA) (Metabolism and nutrition disorders) | 1
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTRAOCULAR (Musculoskeletal and connective tissue disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
HYPOTENSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=11)
BLOOD/BONE MARROW - OTHER (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (Blood and lymphatic system disorders) | 2
CARDIAC ARRHYTHMIA - OTHER (Cardiac disorders) | 1
CARDIAC GENERAL - OTHER (Cardiac disorders) | 1
PAIN - CARDIAC/HEART (Cardiac disorders) | 1
VISION-BLURRED VISION (Eye disorders) | 1
DIARRHEA (Gastrointestinal disorders) | 4
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 2
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Gastrointestinal disorders) | 2
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ORAL CAVITY (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
EDEMA: LIMB (General disorders) | 1
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 5
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2
PAIN - OTHER (General disorders) | 1
RIGORS/CHILLS (General disorders) | 1
SWEATING (DIAPHORESIS) (General disorders) | 1
ALLERGY/IMMUNOLOGY - OTHER (Immune system disorders) | 1
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 1
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Injury, poisoning and procedural complications) | 1
METABOLIC/LABORATORY - OTHER (Investigations) | 1
PLATELETS (Investigations) | 1
WEIGHT LOSS (Investigations) | 1
ANOREXIA (Metabolism and nutrition disorders) | 2
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Metabolism and nutrition disorders) | 2
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Metabolism and nutrition disorders) | 1
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Metabolism and nutrition disorders) | 2
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 3
FRACTURE (Musculoskeletal and connective tissue disorders) | 1
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTRAOCULAR (Musculoskeletal and connective tissue disorders) | 1
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 1
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 1
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 1
PAIN - NECK (Musculoskeletal and connective tissue disorders) | 1
DIZZINESS (Nervous system disorders) | 2
MOOD ALTERATION - AGITATION (Nervous system disorders) | 1
MOOD ALTERATION - ANXIETY (Nervous system disorders) | 1
NEUROLOGY - OTHER (Nervous system disorders) | 2
PAIN - HEAD/HEADACHE (Nervous system disorders) | 2
SEIZURE (Nervous system disorders) | 1
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 1
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 4
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 5
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 1
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 1
HYPOTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes